CLINICAL TRIAL: NCT06036615
Title: The Effect of Exercise Training Intervention and Detraining on Frailty and Fall Risk in Patients With Chronic Heart Failure.
Brief Title: The Effect of Exercise Training and Detraining on Frailty and Fall Risk in Patients With Chronic Heart Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 110/2022
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Chronic Heart Failure
Keywords: Chronic Heart Failure; Cardiac Rehabilitation; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Exercise Group, 6- month combined aerobic, strengthening, mobility- flexibility exercise intervention, 3- month de-training period
  Interventions: Other: Exercise Intervention
- Group B (No Intervention): Control Group, 10- month normal physical activity, without participating in organized sports activities, no intervention

INTERVENTIONS:
Other: Exercise Intervention — Patients that will be randomly assigned to this group will be invited to attend up to 72 exercise sessions (3 sessions per week) for 24 weeks (6 months) following a combined aerobic, strengthening and mobility-flexibility exercise program. After the exercise intervention, the will follow a 3-month de-training period, continuing their normal physical activity.
  Arms: Group A

SUMMARY:
Chronic Heart Failure (CHF) is the endpoint for some cardiac and respiratory conditions as well as ageing affecting 1-2% of the global adult population. CHF requires a costly treatment, frequent hospitalizations due its severe complications leading CHF eventually to a frequent cause of morbidity and mortality worldwide. Another common complication of CHF is frailty. Frailty is a complex clinical syndrome associated with CHF, resulting from multiple organ impairment; physiological reserves decrease and vulnerability to stressors increase. Up to 79% of PwCHF are frail leading to reduced functional capacity, quality of life (QoL), and psychological well-being in CHF, and it is an independent predictor of mortality in cardiovascular disease.

The role of cardiac rehabilitation (CR) programs for PwCHF in preventing frailty has recently draw the attention of the scientific world. Exercise constitutes a unique effective and feasible non-pharmacological treatment for frailty in CHF as it offers such benefits that are irreplaceable by medical treatment, with no side effects, and cost-effective treatment. However, there are no studies examining the effect of training and detraining on muscle strength and balance, fall prevention and fear of falling in PwCHF.

The aim of this randomized controlled trial is to examine whether a 6-month combined aerobic, strengthening and flexibility-mobility CR program and a 3-month de-training period will affect frailty and fall risk in PwCHF. One hundred participants will be randomly allocated into two groups: Group A (Exercise Group) will receive 3 sessions per week for 6 months and Group B(Control Group) will continue their usual physical activity, without participating in organized exercise programs.After the intervention for Group A' will follow a 3- month de-training period and Group B' will continue their normal physical activity. Prior to the group random allocation, part of our assessments at baseline and after 6 (Evaluation A') and 10 months (Evaluation B'), will include demographics and clinical history, physical examination, ECG and echocardiogram, patients' ability to perform daily activities, functional tests, static balance tests, body composition analysis and 24-h heart rhythm holter monitoring. Moreover, we will use questionnaires assessing the QoL of people with CHF, depression, anxiety, sleep quality, cognitive function, fear of falling, physical activity, and sedentary behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs. of either gender
* Confirmed diagnosis (by echocardiography) of HF reduced or preserved left ventricular ejection fraction (HFrEF/ΗFpEF)
* Symptomatic New York Heart Association (NYHA) class II-III

Exclusion Criteria:

* Acute Myocardial Infarction (<4 weeks)
* Severe valvular diseases
* Potentially malignant arrhythmias
* Νeurological, or orthopedic limitations/non- ambulant status
* Cognitive disorders
* Poor regulation of comorbidities
* Already participating in organized exercise programs
* Current pregnancy
* NYHA function class IV
* Inability/unwillingness to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Systolic Function | Baseline
  Evaluation of Left Ventricular Ejection Fraction
Left Ventricular Systolic Function | Evaluation A', 6- months
  Evaluation of Left Ventricular Ejection Fraction
Left Ventricular Systolic Function | Evaluation B', 3 months after evaluation A'
  Evaluation of Left Ventricular Ejection Fraction
Cardiac Autonomic Nervous System Function | Baseline
  Evaluation of Cardiac Autonomic Nervous System Function through 24-h Heart Rhythm Holter Monitor measurement
Cardiac Autonomic Nervous System Function | Evaluation A', 6- months
  Evaluation of Cardiac Autonomic Nervous System Function through 24-h Heart Rhythm Holter Monitor measurement
Cardiac Autonomic Nervous System Function | Evaluation B', 3 months
  Evaluation of Cardiac Autonomic Nervous System Function through 24-h Heart Rhythm Holter Monitor measurement
Body Composition Analysis | Baseline
  Evaluation of Body Composition Analysis
Body Composition Analysis | Evaluation A', 3- months
  Evaluation of Body Composition Analysis
Body Composition Analysis | Evaluation B', 3 months after evaluation A'
  Evaluation of Body Composition Analysis
Six- Minute Walking Test | Baseline
  Estimation of aerobic capacity through six minutes walking test
Six- Minute Walking Test | Evaluation A', 6- months
  Estimation of aerobic capacity through six minutes walking test
Six- Minute Walking Test | Evaluation B', 3 months after evaluation A'
  Estimation of aerobic capacity through six minutes walking test
Timed- Up-and-Go Test | Baseline
  Evaluation of functional capacity using Timed- Up-and-Go Test
Timed- Up-and-Go Test | Evaluation A', 6- months
  Evaluation of functional capacity using Timed- Up-and-Go Test
Timed- Up-and-Go Test | Evaluation B', 3 months after evaluation A'
  Evaluation of functional capacity and mobility using Timed- Up-and-Go Test
4m-Walking Test | Baseline
  Evaluation of functional capacity and mobility using 4m-Walking Test
4m-Walking Test | Evaluation A', 6- months
  Evaluation of functional capacity and mobility using 4m-Walking Test
4m-Walking Test | Evaluation B', 3 months after evaluation A'
  Evaluation of functional capacity and mobility using 4m-Walking Test
30-second Sit-to-Stand (STS)Test | Baseline
  Evaluation of functional capacity and mobility using 30-second STS
30-second Sit-to-Stand (STS)Test | Evaluation A', 6- months
  Evaluation of functional capacity and mobility using 30-second STS
30-second Sit-to-Stand (STS)Test | Evaluation B', 3 months after evaluation A'
  Evaluation of functional capacity and mobility using 30-second STS
5 Sit-to-Stand (5-STS)Test | Baseline
  Evaluation of functional capacity and mobility using 5 Sit-to-Stand
5 Sit-to-Stand (5-STS)Test | Evaluation A', 6- months
  Evaluation of functional capacity and mobility using 5 Sit-to-Stand
5 Sit-to-Stand (5-STS)Test | Evaluation B', 3 months after evaluation A'
  Evaluation of functional capacity and mobility using 5 Sit-to-Stand
mini-BEST Balance Test | Baseline
  Evaluation of balance using mini-BEST Balance Test
mini-BEST Balance Test | Evaluation A', 6- months
  Evaluation of balance using mini-BEST Balance Test
mini-BEST Balance Test | Evaluation B', 3 months after evaluation A'
  Evaluation of balance using mini-BEST Balance Test
Berg Balance Scale Test | Baseline
  Evaluation of balance using Berg Balance Scale Test
Berg Balance Scale Test | Evaluation A', 6- months
  Evaluation of balance using Berg Balance Scale Test
Berg Balance Scale Test | Evaluation B', 3 months after evaluation A'
  Evaluation of balance using Berg Balance Scale Test
Functional Gait Assessment Test | Baseline
  Evaluation of Functional Gait using Functional Gait Assessement Test
Functional Gait Assessment Test | Evaluation A', 6- months
  Evaluation of Functional Gait using Functional Gait Assessement Test
Functional Gait Assessment Test | Evaluation B', 3 months after evaluation A'
  Evaluation of Functional Gait using Functional Gait Assessement Test
Static Balance Test using 3D Balance Force Plate | Baseline
  Evaluation of Static Balance Test using 3D Balance Force Plate
Static Balance Test using 3D Balance Force Plate | Evaluation A', 6- months
  Evaluation of Static Balance Test using 3D Balance Force Plate
Static Balance Test using 3D Balance Force Plate | Evaluation B', 3 months after evaluation A'
  Evaluation of Static Balance Test using 3D Balance Force Plate
Handgrip Strength | Baseline
  Evaluation of Handgrip Strength
Handgrip Strength | Evaluation A', 6- months
  Evaluation of Handgrip Strength
Handgrip Strength | Evaluation B', 3 months after evaluation A'
  Evaluation of Handgrip Strength
Strength of Upper and Lower Extremities | Baseline
  Evaluation of Strength of Upper and Lower Extremities
Strength of Upper and Lower Extremities | Evaluation A', 6- months
  Evaluation of Strength of Upper and Lower Extremities
Strength of Upper and Lower Extremities | Evaluation B', 3 months after evaluation A'
  Evaluation of Strength of Upper and Lower Extremities
Isometric Pulling in a Semi-Squat Position | Baseline
  Evaluation of Isometric Pulling in a Semi-Squat Position
Isometric Pulling in a Semi-Squat Position | Evaluation A', 6- months
  Evaluation of Isometric Pulling in a Semi-Squat Position
Isometric Pulling in a Semi-Squat Position | Evaluation B', 3 months after evaluation A'
  Evaluation of Isometric Pulling in a Semi-Squat Position
30- second Arm Curl Test | Baseline
  Evaluation using Arm Curl Test
30- second Arm Curl Test | Evaluation A', 6- months
  Evaluation using Arm Curl Test
30- second Arm Curl Test | Evaluation B', 3 months after evaluation A'
  Evaluation using Arm Curl Test
Sit-and-Reach Test | Baseline
  Evaluation of mobility-flexibility using Sit-and-Reach Test
Sit-and-Reach Test | Evaluation A', 6- months
  Evaluation of mobility-flexibility using Sit-and-Reach Test
Sit-and-Reach Test | Evaluation B', 3 months after evaluation A'
  Evaluation of mobility-flexibility using Sit-and-Reach Test
Back Scratch Test | Baseline
  Evaluation of mobility using Back Scratch Test
Back Scratch Test | Evaluation A', 6- months
  Evaluation of mobility using Back Scratch Test
Back Scratch Test | Evaluation B', 3 months after evaluation A'
  Evaluation of mobility using Back Scratch Test
SF-36 | Baseline
  Assessment of Quality of Life using SF-36
SF-36 | Evaluation A', 6- months
  Assessment of Quality of Life using SF-36
SF-36 | Evaluation B', 3 months after evaluation A'
  Assessment of Quality of Life using SF-36
I-PAQ | Baseline
  Assessment of Physical Activity using I-PAQ
I-PAQ | Evaluation A', 6- months
  Assessment of Physical Activity using I-PAQ
I-PAQ | Evaluation B', 3 months after evaluation A'
  Assessment of Physical Activity using I-PAQ
Beck Depression Inventory | Baseline
  Assessment of Depression using Beck Depression Inventory
Beck Depression Inventory | Evaluation A', 6- months
  Assessment of Depression using Beck Depression Inventory
Beck Depression Inventory | Evaluation B', 3 months after evaluation A'
  Assessment of Depression using Beck Depression Inventory
Falls Efficacy Scale (FES-I) | Baseline
  Assessment of fear of falling using Falls Efficacy Scale
Falls Efficacy Scale (FES-I) | Evaluation A', 6- months
  Evaluation of fear of falling using Falls Efficacy Scale
Falls Efficacy Scale (FES-I) | Evaluation B', 3 months after evaluation A'
  Assessment of fear of falling using Falls Efficacy Scale
Activities-specific Balance Confidence (ABC) Scale | Baseline
  Assessment of Balance Confidence using ABC
Activities-specific Balance Confidence (ABC) Scale | Evaluation A', 6- months
  Assessment of Balance Confidence using ABC
Activities-specific Balance Confidence (ABC) Scale | Evaluation B', 3 months after evaluation A'
  Assessment of Balance Confidence using ABC
Minnesota Living with Heart Failure (MLHFQ) | Baseline
  Assessment of health-related quality of life using MLHFQ
Minnesota Living with Heart Failure (MLHFQ) | Evaluation A', 6- months
  Assessment of health-related quality of life using MLHFQ
Minnesota Living with Heart Failure (MLHFQ) | Evaluation B', 3 months after evaluation A'
  Assessment of health-related quality of life using MLHFQ
Pittsburgh Sleep Quality Index (PSQI) | Baseline
  Assessment of Sleep Quality using PSQI
Pittsburgh Sleep Quality Index (PSQI) | Evaluation A', 6- months
  Assessment of Sleep Quality using PSQI
Pittsburgh Sleep Quality Index (PSQI) | Evaluation B', 3 months after evaluation A'
  Assessment of Sleep Quality using PSQI
Intrinsic Motivation Inventory (IMI) | Baseline
  Assessment of Intrinsic Motivation using IMI
Intrinsic Motivation Inventory (IMI) | Evaluation A', 6- months
  Assessment of Intrinsic Motivation using IMI
Intrinsic Motivation Inventory (IMI) | Evaluation B', 3 months after evaluation A'
  Assessment of Intrinsic Motivation using IMI
Hamilton Rating Scale for Depression (HRSD) and Hamilton Anxiety Rating Scale (HARS) | Baseline
  Assessment of Depression and Anxiety using HRSD and HARS
Hamilton Rating Scale for Depression (HRSD) and Hamilton Anxiety Rating Scale (HARS) | Evaluation A', 6- months
  Assessment of Depression and Anxiety using HRSD and HARS
Hamilton Rating Scale for Depression (HRSD) and Hamilton Anxiety Rating Scale (HARS) | Evaluation B', 3 months after evaluation A'
  Assessment of Depression and Anxiety using HRSD and HARS
Montreal Cognitive Assessment Test (MOCA) | Baseline
  Assessment of cognitive function using MOCA
Montreal Cognitive Assessment Test (MOCA) | Evaluation A', 6- months
  Assessment of cognitive function using MOCA
Montreal Cognitive Assessment Test (MOCA) | Evaluation B', 3 months after evaluation A'
  Assessment of cognitive function using MOCA
Falls | Baseline
  Assessment of the number of weekly falls
Falls | Evaluation A', 6- months
  Assessment of the number of weekly falls
Falls | Evaluation B', 3 months after evaluation A'
  Assessment of the number of weekly falls
Evaluation of Physical Activity and Sleep Quality using a wearable device | Baseline
  Evaluation of Physical Activity and Sleep Quality using a wearable device
Evaluation of Physical Activity and Sleep Quality using a wearable device | Evaluation A', 6- months
  Evaluation of Physical Activity and Sleep Quality using a wearable device
Evaluation of Physical Activity and Sleep Quality using a wearable device | Evaluation B', 3 months after evaluation A'
  Evaluation of Physical Activity and Sleep Quality using a wearable device
Foot Preference Questionnaire (FPQ) | Baseline
  Assessment of Foot Preference during static balance or activities using FPQ
Foot Preference Questionnaire (FPQ) | Evaluation A', 6- months
  Assessment of Foot Preference during static balance or activities using FPQ
Foot Preference Questionnaire (FPQ) | Evaluation B', 3 months after evaluation A'
  Assessment of Foot Preference during static balance or activities using FPQ
Fear of Falling and Activity Restriction (SAFE) | Baseline
  Assessement of Fear of Falling and Activity Restriction (SAFE)
Fear of Falling and Activity Restriction (SAFE) | Evaluation A', 6- months
  Assessment of Fear of Falling and Activity Restriction (SAFE)
Fear of Falling and Activity Restriction (SAFE) | Evaluation B', 3 months after evaluation A'
  Assessment of Fear of Falling and Activity Restriction (SAFE)
Trail Making Test | Baseline
  Assessment of visual attention and task switching using Trail Making Test
Trail Making Test | Evaluation A', 6- months
  Assessment of visual attention and task switching using Trail Making Test
Trail Making Test | Evaluation B', 3 months after evaluation A'
  Assessment of visual attention and task switching using Trail Making Test

CONTACTS AND LOCATIONS:
Overall Officials: Evangelia Kouidi, Professor, Study Chair — Director of Sports Medicine Laboratory, Aristotle University of Thessaloniki, Greece
Locations (1):
- Sports Medicine Laboratory, Aristotle University of Thessaloniki, Thessaloniki, Thermi, Greece